CLINICAL TRIAL: NCT00834860
Title: The Response and Outcomes of Pegylated Interferon Plus Ribavirin Combination Therapy for Chronic Hepatitis C Patients Concomitant With Hepatocellular Carcinoma
Brief Title: Peginterferon Plus Ribavirin for Hepatitis C Patients Concomitant With Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Wan-Long Chuang, MD., Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUH-IRB-960043
Record Dates: First submitted 2009-02-01; First posted 2009-02-03 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2009-02

CONDITIONS: Chronic Hepatitis C; Hepatocellular Carcinoma
Keywords: chronic hepatitis C; sustained virological response; peginterferon; ribavirin; neoplasm
MeSH Terms: conditions — Hepatitis C, Chronic; Carcinoma, Hepatocellular; Neoplasms | interventions — Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CHC, HCC (Active Comparator): 100 naïve CHC patients concomitant with hepatocellular carcinoma without clinical evidence of HCC recurrence more than 3 months after curative treatments.
  Interventions: Drug: peginterferon alpha-2a and ribavirin
- CHC, LC (Active Comparator): 100 naïve CHC patients without malignancy
  Interventions: Drug: peginterferon alpha-2a and ribavirin

INTERVENTIONS:
Drug: peginterferon alpha-2a and ribavirin — They received peginterferon alpha-2a (180 μg/week) and weight-based ribavirin 1000-1200 mg/day, with a 24-week follow-up period.
  Other Names: Pegasys and Robatrol

SUMMARY:
Combination therapy with pegylated interferon-alpha plus ribavirin has greatly improved the treatment efficacy and is the mainstream of treatment for chronic hepatitis C infection. The efficacy and safety of pegylated interferon-alpha plus ribavirin combination therapy and its impact on the outcome in chronic hepatitis C patients concomitant with hepatocellular carcinoma deserve to be elucidated.

The purposes of this study are:

1. To evaluate the efficacy and safety of pegylated interferon-alpha 2a plus ribavirin combination therapy in chronic hepatitis C patients concomitant with hepatocellular carcinoma.
2. To investigate the role of baseline and on-treatment factors on the response to pegylated interferon-alpha 2a plus ribavirin combination therapy in chronic hepatitis C patients concomitant with hepatocellular carcinoma.

DETAILED DESCRIPTION:
A prospective, hospital-based study enrolling 100 chronic hepatitis C patients concomitant with hepatocellular carcinoma and other sex- and age-matched 100 chronic hepatitis C patients without malignancy will be conducted. The 100 chronic hepatitis C patients concomitant with hepatocellular carcinoma will receive pegylated interferon-alpha 2a plus ribavirin combination therapy at remission phase after oncological treatments and/or interventions. The other 100 chronic hepatitis C patients without malignancy receiving the same antiviral therapy will serve as controls. The primary outcome measurement is sustained virological response and safety, whilst the secondary measurement is rapid virological and early virological response.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients >18 years of age
* Histopathological diagnosis of hepatocellular carcinoma >3 months before entry (Arm A)
* Received curative therapies, including surgery, ablation therapy or liver transplantation >3 months before entry (ArmA)
* No evidence of hepatocellular carcinoma by imaging or histopathological studies at entry
* Patients have never been treated with traditional interferon plus ribavirin or peginterferon plus ribavirin
* Serologic evidence of chronic hepatitis C infection by an anti-HCV antibody test
* Detectable serum HCV-RNA
* Liver biopsy findings consistent with the diagnosis of chronic hepatitis C infection with or without compensated cirrhosis (Exception: hemophiliacs in whom biopsy is medically contra-indicated do not require biopsy.)
* Compensated liver disease (Child-Pugh Grade A clinical classification)
* Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug
* All fertile males and females receiving ribavirin must be using two forms of effective contraception during treatment and during the 6 months after treatment end

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding
* Present therapy with any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) within 6 months prior to the first dose of study drug
* Any investigational drug 6 weeks prior to the first dose of study drug
* Co-infection with active hepatitis A, hepatitis B and/or human immunodeficiency virus (HIV)
* History or other evidence of a medical condition associated with chronic liver disease other than HCV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* Clinical evidence of hepatocellular carcinoma
* History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
* Neutrophil count <1500 cells/mm3 or platelet count <90,000 cells/mm3 at screening
* Serum creatinine level >1.5 times the upper limit of normal at screening
* History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease
* History of a severe seizure disorder or current anticonvulsant use
* History of immunologically mediated disease, chronic pulmonary disease associated with functional limitation, severe cardiac disease, major organ transplantation or other evidence of severe illness, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* History of thyroid disease poorly controlled on prescribed medications, elevated thyroid stimulating hormone (TSH) concentrations with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease
* Evidence of severe retinopathy (e.g. CMV retinitis, macula degeneration)
* Evidence of drug abuse (including excessive alcohol consumption>40 g/day) within one year of study entry
* Inability or unwillingness to provide informed consent or abide by the requirements of the study
* Male partners of women who are pregnant
* Hgb <11 g/dL in women or <12 g/dL in men at screening
* Any patient with major thalassemia
* Patients with documented or presumed coronary artery disease or cerebrovascular disease should not be enrolled if, in the judgment of the investigator, an acute decrease in hemoglobin by up to 4 g/dL (as may be seen with ribavirin therapy) would not be well-tolerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Efficacy: sustained virological response (SVR), HCV RNA seronegative by PCR throughout 24-week off-treatment period. | 1.5 years

SECONDARY OUTCOMES:
Rapid virologic response (RVR), HCV RNA seronegative by PCR at week 4. | 1.5 years
Early virological response (EVR), by PCR-negative or at least 2 logs decline from baseline of serum HCV RNA at 12 weeks of treatment. | 1.5 years
Safety: adverse event rate and profile. | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Long Chuang, MD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Lauer GM, Walker BD. Hepatitis C virus infection. N Engl J Med. 2001 Jul 5;345(1):41-52. doi: 10.1056/NEJM200107053450107. No abstract available. PMID 11439948
- [Background] Chuang WL, Chang WY, Lu SN, Su WP, Lin ZY, Chen SC, Hsieh MY, Wang LY, You SL, Chen CJ. The role of hepatitis B and C viruses in hepatocellular carcinoma in a hepatitis B endemic area. A case-control study. Cancer. 1992 Apr 15;69(8):2052-4. doi: 10.1002/1097-0142(19920415)69:83.0.co;2-n. PMID 1311978
- [Background] Chuang WL, Yu ML, Dai CY, Chang WY. Treatment of chronic hepatitis C in southern Taiwan. Intervirology. 2006;49(1-2):99-106. doi: 10.1159/000087271. PMID 16166797
- [Background] Yu ML, Dai CY, Chen SC, Lee LP, Huang JF, Lin ZY, Hsieh MY, Wang LY, Chuang WL, Chang WY. A prospective study on treatment of chronic hepatitis C with tailored and extended interferon-alpha regimens according to pretreatment virological factors. Antiviral Res. 2004 Jul;63(1):25-32. doi: 10.1016/j.antiviral.2004.01.002. PMID 15196817
- [Background] McHutchison JG, Gordon SC, Schiff ER, Shiffman ML, Lee WM, Rustgi VK, Goodman ZD, Ling MH, Cort S, Albrecht JK. Interferon alfa-2b alone or in combination with ribavirin as initial treatment for chronic hepatitis C. Hepatitis Interventional Therapy Group. N Engl J Med. 1998 Nov 19;339(21):1485-92. doi: 10.1056/NEJM199811193392101. PMID 9819446
- [Background] Fried MW, Shiffman ML, Reddy KR, Smith C, Marinos G, Goncales FL Jr, Haussinger D, Diago M, Carosi G, Dhumeaux D, Craxi A, Lin A, Hoffman J, Yu J. Peginterferon alfa-2a plus ribavirin for chronic hepatitis C virus infection. N Engl J Med. 2002 Sep 26;347(13):975-82. doi: 10.1056/NEJMoa020047. PMID 12324553
- [Background] Chuang WL, Dai CY, Chen SC, Lee LP, Lin ZY, Hsieh MY, Wang LY, Yu ML, Chang WY. Randomized trial of three different regimens for 24 weeks for re-treatment of chronic hepatitis C patients who failed to respond to interferon-alpha monotherapy in Taiwan. Liver Int. 2004 Dec;24(6):595-602. doi: 10.1111/j.1478-3231.2004.0954.x. PMID 15566510
- [Background] Yu ML, Lin SM, Chuang WL, Dai CY, Wang JH, Lu SN, Sheen IS, Chang WY, Lee CM, Liaw YF. A sustained virological response to interferon or interferon/ribavirin reduces hepatocellular carcinoma and improves survival in chronic hepatitis C: a nationwide, multicentre study in Taiwan. Antivir Ther. 2006;11(8):985-94. PMID 17302368
- [Background] Huang JF, Yu ML, Lee CM, Dai CY, Hou NJ, Hsieh MY, Wang JH, Lu SN, Sheen IS, Lin SM, Chuang WL, Liaw YF. Sustained virological response to interferon reduces cirrhosis in chronic hepatitis C: a 1,386-patient study from Taiwan. Aliment Pharmacol Ther. 2007 May 1;25(9):1029-37. doi: 10.1111/j.1365-2036.2007.03297.x. PMID 17439503
- [Derived] Huang JF, Yeh ML, Yu ML, Dai CY, Huang CF, Huang CI, Tsai PC, Lin PC, Chen YL, Chang WT, Hou NJ, Lin ZY, Chen SC, Chuang WL. The tertiary prevention of hepatocellular carcinoma in chronic hepatitis C patients. J Gastroenterol Hepatol. 2015 Dec;30(12):1768-74. doi: 10.1111/jgh.13012. PMID 26094738